CLINICAL TRIAL: NCT02251249
Title: Impairment of Gastric Emptying During Acute Phase of Myocardial Infarction. Impact on Oral Antiplatelet Treatment Efficacy. The GASTRIM Study.
Acronym: GASTRIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2013/19
Record Dates: First submitted 2014-09-24; First posted 2014-09-29 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Impairment of Gastric Emptying; Acute Phase of Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- STEMI Group (Experimental)
  Interventions: Drug: Paracetamol concentration time curve from 0 to 120 min
- Stable patient Group (Other): Patient referred for angioplasty for angina or non-ST-segment elevation myocardial infarction (NSTEMI)
  Interventions: Drug: Paracetamol concentration time curve from 0 to 120 min

INTERVENTIONS:
Drug: Paracetamol concentration time curve from 0 to 120 min — It consists in oral ingestion of 1.5g of paracetamol (Contents of 3 Doliprane® capsules 500 mg) and 60 mg prasugrel (6 tablets Efient ® 10 mg) or 180 mg ticagrelor ( 2 tablets Brilique ® 90 mg) with water. Then Paracetamol concentration is followed by the realization of the curve of concentration of paracetamol in plasma samples. These samples are taken at 15 min intervals during the first 2 hours.

SUMMARY:
Oral antiplatelet therapy is a key treatment of the STEMI (ST elevation myocardial infarction). Delayed action isn't suitable and has to be elucidated. If a delayed gastric emptying time is observed during STEMI, limiting the use of morphine and encourage the use of prokinetic agents can be a first answer to optimize coronary angioplasty environment.

Investigators propose a study to assess the gastric emptying times at the acute phase of myocardial infarction using a validated paracetamol absorption test. The STEMI group will be compared to in one hand, itself with measures performed 72 hours±12h after the event onset; and on the other hand, to a stable patient group referred for angioplasty for angina or non-ST-segment elevation myocardial infarction (NSTEMI). For STEMI group and stable patient group, the delay of apparition of Prasugrel or Ticagrelor efficacy will be determined by VerifyNow® test and correlated to gastric emptying times.

DETAILED DESCRIPTION:
Oral antiplatelet therapy is a key treatment of the STEMI (ST elevation myocardial infarction). Delayed action isn't suitable and has to be elucidated. If a delayed gastric emptying time is observed during STEMI, limiting the use of morphine and encourage the use of prokinetic agents can be a first answer to optimize coronary angioplasty environment.

Investigators propose a study to assess the gastric emptying times at the acute phase of myocardial infarction using a validated paracetamol absorption test. The STEMI group will be compared to in one hand, itself with measures performed 72 hours±12h after the event onset; and on the other hand, to a stable patient group referred for angioplasty for angina or non-ST-segment elevation myocardial infarction (NSTEMI). For STEMI group and stable patient group, the delay of apparition of Prasugrel or Ticagrelor efficacy will be determined by VerifyNow® test and correlated to gastric emptying times.

Paracetamol absorption test is a safe, cheap and well validated method to assess these times including during the STEMI period. This one consists in oral ingestion of 1.5g of paracetamol followed by the realization of the curve of concentration of paracetamol in plasma samples. These samples are taken at 15 min intervals during the first 2 hours.

In the same time the curve of Platelet reactivity Unit (PRU) obtained by VerifyNow® tests will be determined with the goal to establish a relation between gastric emptying times and delayed observed antiplatelet activity.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years weighing between 65 and 85 Kg
* Referred for STEMI within 6 hours from beginning of chest pain or stable coronary artery disease requiring a loading dose of Prasugrel or Ticagrelor according to the international recommendations.
* No previous treatment with Clopidogrel, Prasugrel or Ticagrelor.
* Patient fasting for at least 6 hours.
* Affiliate or receiving a social security system.
* Written informed consent.

Exclusion Criteria:

* Allergy or contraindication to paracetamol, Prasugrel or Ticagrelor
* Paracetamol ingestion in the previous 48 hours
* Patient treated with drugs supposed to alter gastric emptying times (calcium antagonists, Alimentary tract treatments, opioid analgesics, tricyclic antidepressants, antibiotics).
* Conditions or pathologies supposed to alter gastric emptying times (Thyroid dysfunction, chronic renal failure, Parkinson's disease, scleroderma, amyloidosis, any gastrointestinal disease, any not cured malignancy, and any advanced psychiatric or neurological disease).
* Presence of vomiting
* Cardiogenic shock, ventricular arrhythmia or resuscitated cardiac arrest
* Hepatic insufficiency
* Severe respiratory disease
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2016-09-25 (Actual)

PRIMARY OUTCOMES:
Determination of the paracetamol concentration time curve at the time of STEMI Onset | Every 15 minutes since inclusion (STEMI onset ) up to 120 minutes
  Taking of blood samples every 15 minutes for patients of STEMI Group
Determination of the paracetamol concentration time curve 72 hours after time of STEMI Onset | Every 15 minutes since 72 hours after STEMI onset up to 120 minutes
  Taking of blood samples every 15 minutes for patients of STEMI Group
Determination of the paracetamol concentration time curve for Stable patient Group | Every 15 minutes since inclusion up to 120 minutes
  Taking of blood samples every 15 minutes for Stable patient Group

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux - Hôpital du Haut Lévèque, Pessac, France